CLINICAL TRIAL: NCT02829255
Title: Effect of High Altitude Exposure, Acclimatization and Re-exposure on Cerebral Autoregulation in Lowlanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB15-2709_V4
Record Dates: First submitted 2016-04-01; First posted 2016-07-12 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Effect of High Altitude
Keywords: High altitude; Cerebral autoregulation; Transfer function analysis
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altitude exposure (Experimental): Acute high altitude exposure followed by 8 day acclimatization and reexposure for 8 days after 6 days at low altitude
  Interventions: Other: altitude exposure

INTERVENTIONS:
Other: altitude exposure — altitude exposure

SUMMARY:
Prospective interventional trial in lowlanders evaluating the effect of acute exposure, acclimatization and re-exposure to high altitude on cerebral autoregulation

DETAILED DESCRIPTION:
Baseline measurements will be performed in Santiago de Chile, 520 m, over the course of 3 days. Participants will then travel by commercial airline (5 h flight) and by bus (3 h ride) to the ALMA base camp located at 2900 m near San Pedro de Atacama, northern Chile. Participants will stay there for the next 8 nights and they will be spend the days (6-8 h daily) at the telescope station at 5050 m while undergoing testing as described above at the first and the last day at 5050m. Daily transports from 2900 to 5050 m will be by car (1 h ride, one way). After the first 8 day altitude sojourn participants will return to the Santiago area (520 m) for a 6 day recovery period.

A second altitude sojourn with an identical schedule as the one described above and a final low altitude stay of 3 days will follow.

ELIGIBILITY:
Inclusion Criteria:

* Born, raised and currently living <800m
* No overnight stay at altitudes >1500 m 4 weeks before the study

Exclusion Criteria:

* Previous altitude intolerance to altitude <3000 m
* Pregnancy
* Health impairment, which requires regular treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04-09 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-04 (Actual)

PRIMARY OUTCOMES:
Coherence between middle cerebral artery blood flow velocity and systemic blood pressure as measure of cerebral autoregulation. | day 1; day 2 first cycle
  Change in magnitude of the coefficient of coherence between blood flow velocity in the middle cerebral artery measured by transcranial ultrasound Doppler and systemic blood pressure at day 2 (5050 m) vs. day 1 (520 m) of the first cycle

SECONDARY OUTCOMES:
Coherence between middle cerebral artery blood flow velocity and systemic blood pressure as measure of cerebral autoregulation. | day 1; day 7 first cycle
  Change in magnitude of the coefficient of coherence between blood flow velocity in the middle cerebral artery measured by transcranial ultrasound Doppler and systemic blood pressure at day 7 (5050 m) vs. day 1 (520 m) of the first cycle.
Coherence between middle cerebral artery blood flow velocity and systemic blood pressure as measure of cerebral autoregulation. | day 2; day 7 second cycle
  Change in magnitude of the coefficient of coherence between blood flow velocity in the middle cerebral artery measured by transcranial ultrasound Doppler and systemic blood pressure at day 7 (5050 m) vs. day 2 (5050 m) of the second cycle.
Coherence between middle cerebral artery blood flow velocity and systemic blood pressure as measure of cerebral autoregulation. | day 2 first cycle; day 2 second cycle
  Change in magnitude of the coefficient of coherence between blood flow velocity in the middle cerebral artery measured by transcranial ultrasound Doppler and systemic blood pressure at day 2 (5050 m) second cycle vs. day 2 (5050 m) of the first cycle.
Coherence between middle cerebral artery blood flow velocity and systemic blood pressure as measure of cerebral autoregulation. | day 7 first cycle; day 7 second cycle
  Change in magnitude of the coefficient of coherence between blood flow velocity in the middle cerebral artery measured by transcranial ultrasound Doppler and systemic blood pressure at day 7 (5050 m) second cycle vs. day 7 (5050 m) of the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No